CLINICAL TRIAL: NCT00927966
Title: Phase I Clinical Trial of RAD001 in Combination With CP-751,871 in Patients With Advanced Sarcomas and Other Malignant Neoplasms
Brief Title: RAD001 in Combination With CP-751,871 in Patients Wtih Advanced Sarcomas and Other Malignant Neoplasms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzanne George, MD (Other)
Collaborators: Brigham and Women's Hospital (Other); Novartis (Industry); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Suzanne George, MD, Clinical Director Center for Sarcoma and Bone Oncology, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-091
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Sarcoma; Solid Tumor
Keywords: RAD001; CP-751,871; advanced sarcoma; advanced malignant solid tumor
MeSH Terms: conditions — Sarcoma | interventions — Everolimus; figitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 in combination with figitumumab (Experimental)
  Interventions: Drug: RAD001; Drug: CP-751,871

INTERVENTIONS:
Drug: RAD001 — Taken orally once a day.
Drug: CP-751,871 — Given intravenously on Day 1 of a 21-day cycle

SUMMARY:
The purpose of this research study is to determine the safety of the combination of RAD001 and CP-751,871, as well as the highest dose of this combination that can be given to people safely. RAD001 is a newly discovered drug that may stop cancer cells from growing abnormally. This drug has been extensively studied in many cancers. In particular, it has shown to be effective in slowing down the growth of kidney cancer. CP-751,871 is another newly discovered drug that may stop tumor growth. It is currently being studied in a wide variety of cancers, and information from those other research studies suggests that these two drugs in combination may help to stop cancer growth.

DETAILED DESCRIPTION:
* In this research study, each "cycle" of study drug dosing lasts 21 days. In the first cycle, participants will come to the clinic on Days 1, 8, and 15. During cycles 2 through 4, participants will come to the clinic on Days 1 and 8. The rest of the clinic visits will occur on Day 1 of every cycle thereafter.
* During each cycle, participants will take RAD001 orally, once a day in the morning. In addition, participants will receive CP-751,871 intravenously once every cycle on the first day of each cycle.
* Since we are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects, not everyone who participates in this research study will receive the same dose of the study drug. The dose will depend on the number of participants enrolled in the study and how well they tolerated their doses.
* Participants may remain on this research study as long as they do not have serious side effects or their diseae does not get worse.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced sarcoma or other advanced malignant solid tumor for which no known curative therapy exists. Patients must have had prior progression on, intolerance or refused approved standard therapies proven to prolong life.
* Measurable disease per RECIST. A lesion in a previously irradiated area is eligible to be considered as measurable disease as long as there is objective evidence of progression of the lesion prior to study enrollment
* 18 years of age or older
* ECOG Performance Status 0-1
* Participants must have normal organ and marrow function as outlined in the protocol
* Fully recovered from the acute effects of prior cancer therapy before initiation of study drug
* Negative urine or serum pregnancy test within 7 days prior to initiation of study drug for women of child-bearing potential
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for up to 6 months after the last dose of study drug

Exclusion Criteria:

* Participants with gastrointestinal tumors (GIST) on approved tyrosine kinase inhibitors within 2 weeks prior to study entry
* All other participants who have had systemic anti-cancer therapy within 3 weeks (8 weeks for nitrosoureas or mitomycin C) prior to study entry
* Participants who have had radiotherapy and/or major surgery within 2 weeks prior to study entry
* Concurrent use of any other anti-cancer therapies, study agents, growth hormones, growth hormone inhibitors or aminoglycoside antibiotics
* Participants who have had chronic high dose immunosuppressive steroid therapy within 2 weeks prior to enrollment. Previous high dose steroid treatment > 2 weeks prior to study entry, topical and inhaled corticosteroids are allowed
* Presence of symptomatic or uncontrolled brain or central nervous system metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to RAD001 and/or CP-751,871
* Participants receiving any medications or substances that are inhibitors or inducers of CYP3A
* Uncontrolled diabetes
* Bleeding diathesis or requirement for therapeutic anticoagulation
* Uncontrolled intercurrent illness
* Pregnant or nursing women
* HIV positive individuals on combination anti-retroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of daily oral RAD001, administered in combination with CP-751,871 given as an intravenous infusion in patients with advanced sarcomas and other advanced solid tumors that are incurable with any current modality. | 3 years

SECONDARY OUTCOMES:
To assess the pharmacokinetics of this combination regimen. | 3 years
To allow a preliminary assessment of the anti-tumor effects of this novel drug combination. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne George, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States